CLINICAL TRIAL: NCT05962892
Title: A Study of Factors Influencing Recurrence After Thermal Ablation of Papillary Thyroid Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR-11-23-009728
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-02

CONDITIONS: Papillary Thyroid Carcinoma; Thermal Ablation
Keywords: Papillary Thyroid Carcinoma; cohort; Thermal Ablation; Recurrence
MeSH Terms: conditions — Thyroid Cancer, Papillary; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Intervention
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
A prospective cohort of papillary thyroid carcinoma(PTC), patients who received thermal ablation in our hospital since February 2023 was established as the study object. Preoperative and postoperative demographic data, ultrasonography, other relevant laboratory tests, and thyroid disease-related scales such as fatigue, depression, and stress were collected. The influencing factors of PTC recurrence were analyzed.

ELIGIBILITY:
Inclusion Criteria:

①≥18 years old; ② Obtain informed consent; ③ Ultrasonography showed that malignant nodules were single, the maximum diameter of nodules was ≤1cm and the distance from the capsule was ≥2mm. ④ no lymph node metastasis or other extra-glandular metastasis in the neck; ⑤ PTC was confirmed by fine needle puncture pathology; ⑥ Patients who do not meet Article 3, who still strongly request thermal ablation while fully informing the patient of the risk of recurrence, and who have been clinically assessed to be technically capable of thermal ablation Exclusion Criteria:① Pregnant or lactating patients; ② Patients with other malignant tumors and not suitable for ablation by clinical evaluation; ③ Patients who cannot tolerate surgery; ④ Patients with cognitive impairment and other conditions who cannot accurately fill in thyroid-related questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically proven PTC underwent ultrasound-guided percutaneous thermal ablation.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
the recurrence of PTC | 1 to 5 years
  the recurrence of PTC during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No